CLINICAL TRIAL: NCT01756196
Title: Prospective Observational Study of Evaluate the Incidence and Types of Systemic Reactions After Spinal Steroid Injections
Brief Title: Incidence of Various Types of Systemic Reactions Related to Spinal Steroid Injection: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Guen Young Lee, Associate Professor, MD, PhD, Seoul National University Bundang Hospital
Other Study IDs: B-1008/016-004
Record Dates: First submitted 2012-12-19; First posted 2012-12-25 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: Incidence and Types of Systemic Reactions Occurring After Spinal Steroid Injection in a Large Population
Keywords: Spinal injection; Steroid; Systemic reaction; Complication; Side effect; Diabetes mellitus; Hypertension; Risk factor
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Steroid Injection: Reactions associated with spinal steroid injection
  Interventions: Drug: Spinal Steroid Injection

INTERVENTIONS:
Drug: Spinal Steroid Injection — Steroid Injection

SUMMARY:
Many systemic reactions occur commonly after spinal steroid injections, especially in patients, and may be associated with underlying disease, such as hypertension and diabetes mellitus, as well as steroid dose and repetition of spinal steroid injection.

DETAILED DESCRIPTION:
Evaluate the incidence and types of systemic reactions after spinal steroid injections and to investigate the association of spinal steroid injection with patient demographics, history of previous injections, type and dose of steroid, and method and site of previous and current injections.

ELIGIBILITY:
Inclusion Criteria:

* Indicaion of steroid injction.

Exclusion Criteria:

* Contraindiation of steroid injction.

Ages: 13 Years to 94 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving the injection were informed of the aim and protocol of this study and the possible local and systemic reactions associated with spinal steroid injection
Sampling Method: Non-Probability Sample
Enrollment: 997 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
episodes of systemic reactions after spinal steroid injection | 2 weeks
  Evaluation of episodes of systemic reactions after spinal steroid injection

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seoung Nam, Bundang, South Korea

REFERENCES:
- [Result] Goldstein G, Schlesinger DH. Thymopoietin and myasthenia gravis: neostigmine-responsive neuromuscular block produced in mice by a synthetic peptide fragment of thymopoietin. Lancet. 1975 Aug 9;2(7928):256-9. doi: 10.1016/s0140-6736(75)90966-6. PMID 49801